CLINICAL TRIAL: NCT06868901
Title: Evaluation of the 6-month Response Rate According to Two Surgical Techniques (Rotational Atherectomy vs. Angioplasty) to Treat Stenosis of Vascular Accesses in Hemodialysis. A Single-center, Randomized, Single-blind, Superiority-controlled Pilot Study.
Brief Title: Six-month Response Rate According to Two Surgical Techniques (Rotational Atherectomy Versus Angioplasty) to Treat Stenosis of Vascular Accesses in Hemodialysis.
Acronym: ARSAV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NIMAO/2024-1/EF01
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hemodialysis Complication; Dialysis Access Malfunction; Stenosis
Keywords: Arteriovascular fistula; Angioplasty; Balloon; Atherectomy; Fistula; Re-stenosis
MeSH Terms: conditions — Constriction, Pathologic; Fistula | interventions — Atherectomy

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized (ratio 1:1), single-blind (patient), superiority controlled study comparing two surgical techniques for the treatment of restenosis of hemodialysis vascular access: atherectomy + drug-eluting balloon (experimental group "ATH") versus standard angioplasty + drug-eluting balloon (control group "ANG").
  The impact of atherectomy with drug-eluting balloon for the treatment of arteriovenous fistula (AVF) restenosis at 6 months after surgery will be assessed via a comparator group (angioplasty with drug-eluting balloon) and on the basis of a specific judgement criterion, i.e. the occurrence of re-stenosis at this time.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient is blinded to his or her group. The ultrasonographer performing the echodoppler examinations is blinded to the patient's home group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (ANG) (Active Comparator): Treatment of re-stenosis of hemodialysis vascular access using the standard angioplasty + drug-eluting balloon technique.
  Interventions: Procedure: Standard angioplasty + drug-eluting balloon technique
- Experimental group (ATH) (Active Comparator): Treatment of re-stenosis of hemodialysis vascular access using the atherectomy + drug-eluting balloon technique.
  Interventions: Procedure: Atherectomy + drug-eluting balloon

INTERVENTIONS:
Procedure: Standard angioplasty + drug-eluting balloon technique — Treatment of restenosis of hemodialysis vascular access via the standard angioplasty + drug-eluting balloon technique
  Arms: Control group (ANG)
Procedure: Atherectomy + drug-eluting balloon — Treatment of restenosis of hemodialysis vascular access via the atherectomy + drug-eluting balloon technique
  Arms: Experimental group (ATH)

SUMMARY:
A well-functioning hemodialysis vascular access is a decisive factor in the survival of hemodialysis patients, who have a high mortality rate. 85% of these hemodialysis patients, are treated via an arteriovenous fistula (AVF). However, the primary patency of AVFs at 1 year is 60%, mainly due to neointimal hyperplasia developing in the drainage vein, which leads to stenosis and, if left untreated, thrombosis of the AVF. Indeed, forty percent of hemodialysis patients require re-intervention on their vascular access within the year, due to stenosis on their AVF.

Transluminal angioplasty (TLA) is currently used as first-line treatment for these stenoses but TLA itself causes vascular damage, with early recurrence of the stenosis in 50% of cases at 6 months, and necessitating repeated interventions.

In recent years several endovascular techniques have been developed to limit the risk of re-stenosis, none of which have produced significantly better results than simple TLA. Eliminating intimal hyperplasia using a minimally invasive endovascular technique, rather than crushing it with simple angioplasty, would improve restenosis-free survival in these patients.

Today, endovascular rotational atherectomy techniques are available to improve the patency of angioplasty in the treatment of complex arterial lesions of the coronary arteries and lower limbs. The atherotome is a guide-mounted catheter with a small burr at its distal end, which resects the atheromatous plaque whereas angioplasty simply crushes it. Atherectomy is followed by drug-eluting balloon (DEB) angioplasty with paclitaxel release to limit restenosis through its anti-inflammatory and anti-proliferative activity. A few cases of rotational atherectomy for the treatment of calcified stenoses in saphenous vein coronary bypasses have been reported in the literature, with encouraging results. If AVF re-stenosis should occur, the intimal hyperplasia can be removed endovascularly, thereby limiting the risk of short-term iterative stenosis.

The aim of this study was to compare the 6-month re-stenosis rate with this technique (atherectomy + drug-eluting balloon) versus standard angioplasty + drug-eluting balloon for the treatment of restenosis of hemodialysis vascular accesses.

DETAILED DESCRIPTION:
A well-functioning hemodialysis vascular access is a decisive factor in the survival of hemodialysis patients, who have a high mortality rate. 85% of these hemodialysis patients, are treated via an arteriovenous fistula (AVF), which is currently the access offering the best results in terms of patency and infectious risk. However, the primary patency of AVFs at 1 year is 60%, mainly due to the development of neointimal hyperplasia in the drainage vein, which leads to stenosis and, if left untreated, thrombosis of the AVF. Forty percent of hemodialysis patients on AVF will therefore have at least one intervention on their vascular access within the year, due to stenosis on their AVF.

Transluminal angioplasty (TLA) is currently used as first-line treatment for these stenoses. However, TLA itself causes vascular damage, with migration and myofibroblast proliferation responsible for abnormal vascular remodeling, leading to early recurrence of the stenosis in 50% of cases at 6 months, limiting the long-term functionality of these angioplasties and necessitating repeated interventions on these patients. For all these reasons, developing techniques to limit the risk of re-stenosis of hemodialysis AVFs is a public health issue.

In recent years several endovascular techniques have been developed to limit the risk of re-stenosis: paclitaxel-coated "active" balloon angioplasty, bare or covered stenting, none of which have produced significantly better results than simple TLA. Eliminating intimal hyperplasia using a minimally invasive endovascular technique, rather than crushing it with simple angioplasty, would improve restenosis-free survival in these patients, without increasing the burden of management.

Today, endovascular rotational atherectomy techniques are available to improve the patency of angioplasty in the treatment of complex arterial lesions of the coronary arteries and lower limbs. The atherotome is a guide-mounted catheter with a small burr at its distal end, which resects the atheromatous plaque where angioplasty simply crushes it. Atherectomy is followed by drug-eluting balloon angioplasty with paclitaxel release to limit restenosis through its anti-inflammatory and anti-proliferative activity. A few cases of rotational atherectomy for the treatment of calcified stenoses in saphenous vein coronary bypasses have been reported in the literature, with encouraging results and the absence of complications, notably perforation. If AVF re-stenosis should occur, the intimal hyperplasia can be removed endovascularly, thereby limiting the risk of short-term iterative stenosis.

The aim of this study was to compare the 6-month re-stenosis rate with this technique (atherectomy + drug-eluting balloon) versus standard angioplasty + drug-eluting balloon for the treatment of restenosis of hemodialysis vascular accesses.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient on arteriovenous fistula (AVF) with re-stenosis defined on echodoppler by a combination of >50% venous lumen reduction with a systolic peak ratio >2 associated with either : i) an internal residual diameter of < 2 mm, or ii) a flow reduction > 25% or a flow rate < 500 ml/min.
* Patient with at least one history of angioplasty on his/her AVF at the same site.
* Patient available for 6-month follow-up.
* Patient with free and informed consent and signed consent form.
* Patient affiliated with or benefiting from a health insurance plan.

Exclusion Criteria:

* Patient with an intraoperative technical impossibility.
* Patient with a septic complication.
* Patient participating in another interventional trial.
* Patient in an exclusion period determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Patient for whom it is impossible to give informed information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Re-stenosis rate at 6 months in the control group | At 6 months postoperative
  YES/NO Significant restenosis is defined on echodoppler by a combination of > 50% venous lumen reduction with a systolic peak ratio > 2 associated with: i) either an internal residual diameter < 2 mm, ii) or a flow reduction > 25% or flow < 500 ml/min.
Re-stenosis rate at 6 months in the experimental group | At 6 months postoperative
  YES/NO Significant restenosis is defined on echodoppler by a combination of > 50% venous lumen reduction with a systolic peak ratio > 2 associated with: i) either an internal residual diameter < 2 mm, ii) or a flow reduction > 25% or flow < 500 ml/min.

SECONDARY OUTCOMES:
Time to re-stenosis in the control group | Up to 6 months postoperative
  Time (days) from surgery to onset of restenosis as defined above.
Time to re-stenosis in the experimental group | Up to 6 months postoperative
  Time (days) from surgery to onset of restenosis as defined above.
Rate of complications in the control group | Up to 6 months' follow-up.
  Collection of complications related to surgical technique: perforation (assessed by the operator intraoperatively: extravasation of contrast medium at fistulographic control), false aneurysm (assessed at follow-up echodoppler).
Rate of complications in the experimental group | Up to 6 months' follow-up.
  Collection of complications related to surgical technique: perforation (assessed by the operator intraoperatively: extravasation of contrast medium at fistulographic control), false aneurysm (assessed at follow-up echodoppler).
Intermediate re-stenosis at 1 month in the control group | At 1 month postoperative
  Intermediate patency assessed by significant restenosis as defined above
Intermediate re-stenosis at 1 month in the experimental group | At 1 month postoperative
  Intermediate patency assessed by significant restenosis as defined above
Intermediate re-stenosis at 3 months in the control group | At 3 months postoperative
  Intermediate patency assessed by significant restenosis as defined above
Intermediate re-stenosis at 3 months in the experimental group | At 3 months postoperative
  Intermediate patency assessed by significant restenosis as defined above
Systolic velocity in the control group | At 3 months postoperative
  Systolic velocity (ml/s) assessed by echodoppler
Systolic velocity in the experimental group | At 3 months postoperative
  Systolic velocity (ml/s) assessed by echodoppler
Systolic velocity in the control group | At 6 months postoperative
  Systolic velocity (ml/s) assessed by echodoppler
Systolic velocity in the experimental group | At 6 months postoperative
  Systolic velocity (ml/s) assessed by echodoppler
Venous lumen at 1 month in the control group | At 1 month postoperative
  Measurement of venous lumen as a percentage on echodoppler
Venous lumen at 1 month in the experimental group | At 1 month postoperative
  Measurement of venous lumen as a percentage on echodoppler
Venous lumen at 3 months in the control group | At 3 months postoperative
  Measurement of venous lumen as a percentage on echodoppler
Venous lumen at 3 months in the experimental group | At 3 months postoperative
  Measurement of venous lumen as a percentage on echodoppler
Venous lumen at 6 months in the control group | At 6 months postoperative
  Measurement of venous lumen as a percentage on echodoppler
Venous lumen at 6 months in the experimental group | At 6 months postoperative
  Measurement of venous lumen as a percentage on echodoppler
Re-intervention rate for thrombosis in the control group | Up to 6 months postoperative
  Occurrence of re-intervention for thrombosis: yes/no.
Re-intervention rate for thrombosis in the experimental group | Up to 6 months postoperative
  Occurrence of re-intervention for thrombosis: yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Elsa FAURE, Dr., Principal Investigator — Vascular and Thoracic Surgery department, Nîmes University Hospital, France

IPD SHARING:
Plan to Share IPD: No
Data is managed by the BESPIM (Biostatistics Epidemiology Public Health & Innovation in Methodology) of the Nîmes University Hospital. The conditions for transferring all or part of the research database are decided by the research sponsor, and will be set out in a written contract.